CLINICAL TRIAL: NCT05307614
Title: A Single Center, Open Label, Randomized, Single-dose, 2 Way Cross-over Study to Explore the Relative Bioavailability of Moksi 400mg (Moxifloxacin) Tablet and Avelox 400mg (Moxifloxacin) Tablet Under Fasting Conditions in Healthy Male Pakistani Subjects
Brief Title: Bioequivalence Study of Moksi® 400mg Tablet and Avelox® 400mg Tablet (Moxifloxacin) Under Fasting Condition in Healthy Adult Pakistani Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MOXI1001; CB-023-MOX-2017/Protocol/2.0 (Other: Center for Bioequivalence Studies and Clinical Research (CRO))
Record Dates: First submitted 2022-03-21; First posted 2022-04-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Bioequivalence
Keywords: Moxifloxacin; Fluoroquinolone; Bioequivalence; Pakistani population
MeSH Terms: interventions — Tablets; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: Cross Over
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moksi® 400mg Tablet of Abbott (Experimental): Healthy subjects were orally administered a single dose of Moksi® 400mg Tablet (Moxifloxacin) under fasting condition
  Interventions: Drug: Moksi® 400mg Tablet; Drug: Drug: Avelox® 400Mg Tablet
- Avelox® 400mg Tablet of Bayer (Active Comparator): Healthy subjects were orally administered a single dose of Avelox® 400mg Tablet (Moxifloxacin) under fasting condition.
  Interventions: Drug: Moksi® 400mg Tablet; Drug: Drug: Avelox® 400Mg Tablet

INTERVENTIONS:
Drug: Moksi® 400mg Tablet — Single dose of Moxifloxacin 400 mg Tablet was administered after a 10-hour overnight fast.
  Other Names: Moksi®
Drug: Drug: Avelox® 400Mg Tablet — Single dose of Moxifloxacin 400 mg Tablet was administered after a 10-hour overnight fast.
  Other Names: Avelox®

SUMMARY:
Single dose, two way crossover Bioequivalence (BE) study to evaluate the comparative bioavailability of moxifloxacin.

DETAILED DESCRIPTION:
A single center, single-dose, open-label randomized , 2-way crossover Bioequivalence study in healthy Pakistani subjects. Study drugs, Moksi® 400 mg (Moxifloxacin) Tablet manufactured by Abbot Laboratories (Pakistan) Limited and Avelox® 400mg (Moxifloxacin) Tablet manufactured by Bayer HealthCare Pharmaceuticals Inc were administered in two periods separated by a washout period of seven (07) days. After dosing, serial blood samples were collected for a period of 72.0 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers aged 18 to 55 years inclusive.
2. Subjects with a body mass index from 18.5 to 30 kg/m2 (both inclusive).
3. Subjects who are healthy as determined by routine physical examination,including vital sign monitoring (ie, blood pressure, heart rate,and temperature), 12 lead ECG ,chest X ray and laboratory analysis (ie, hematology, blood biochemistry and urinalysis), as determined by the investigator.
4. Subjects should have negative urine test for drugs of abuse (Opiates, benzodiazepines, amphetamines, barbiturates, cannabinoids and cocaine will be tested) and alcohol breath analysis at screening and prior to each check-in.
5. Subjects and their partners are willing to use reliable non-hormonal contraceptive methods (condoms, diaphragm, non-hormonal intra- uterine device (IUD), female or male sterilization or sexual abstinence) throughout the study and up to 30 days after the last administration of the study drug
6. All subjects should be free from any epidemic or contagious diseases (e.g. Malaria, Dengue).
7. Subjects will be able to, understand and sign the Informed Consent Form for Medical Screening during their screening visit and Participation Informed Consent Form on study check-In day.

Exclusion Criteria:

1. History of smoking (> 5 cigarette/day), alcoholism, and positive test for drug of abuse, heavy pan or gutka user as judged by teeth / mouth inspection.
2. Subjects with clinically relevant evidence of cardiovascular, gastrointestinal/hepatic, renal, psychiatric, respiratory, urogenital, hematologic/immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/ connective tissue, musculoskeletal, metabolic/nutritional, drug hypersensitivity, allergy, endocrine, major surgery or other relevant diseases as revealed by medical history, physical examination, and laboratory assessments which may interfere with the absorption, distribution, metabolism or elimination of drugs or constitute a risk factor when taking study medication.
3. Subject is allergic to Moxifloxacin and/or other fluoroquinolones
4. Subject has received any investigational drug within four weeks.
5. Subjects with known prolongation of the QT interval.
6. Subjects receiving Class IA (e.g. quinidine, procainamide) or Class III (e.g. amiodarone, sotalol) antiarrhythmic agents.
7. Subjects with salt imbalance in the blood (especially low levels of potassium or magnesium in the blood)
8. Subject taking any vitamins or herbal supplements during within last 14 days of drug administration.
9. Donation or loss of more than 450 mL of blood within 3 months prior to the screening.
10. Ingestion of OTC drug, within 7 days of drug administration (e.g. aspirin, ibuprofen).
11. History of intake of any prescribed medicine during a period of 30 days, prior to drug administration day of study.
12. History of any significant illness in the last four weeks
13. Subjects who smoke and/or take nicotine in any form. Non-smoking subjects, who have previously smoked, should at least be non-smoking for 6 months prior to dosing.
14. Concomitant treatment with systemic ketoconazole, cyclosporine, itraconazole, verapamil and dronedarone.
15. Consumption of grapefruit and/or its products within 14 days prior to the start of study.
16. Subjects who test positive for syphilis (VDRL)or who are known to have serum hepatitis or who are carriers of the Hepatitis B surface antigen (HBs Ag) or are carriers of antibodies to hepatitis C virus (anti-HCV) or to the human immunodeficiency virus (HIV-1 or HIV-2)
17. Individuals having undergone any major surgery within 3 months prior to the start of the study,
18. Subject has a history of any illness that, in the opinion of investigator might confound the result of the study or post additional risk in administrating moxifloxacin to the subject.
19. Inability to take oral medication.
20. Subjects with any condition, which, in the opinion of the Investigator, may interfere with the absorption, distribution, metabolism or elimination of drugs.
21. Subjects with clinically significant abnormalities in investigations (safety assessments) as determined by the Investigator

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 38 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2019-04-23 (Actual); Study Completion 2019-04-27 (Actual)

PRIMARY OUTCOMES:
Cmax | 0-72 hours post dose
  maximum plasma concentration of Moxifloxacin
AUC last (AUC 0-t) | 0-72 hours post dose
  Area under plasma concentration time curve from zero to time of the last measurable concentration
AUC total (AUC 0-∞) | 0-72 hours post dose
  area under the plasma concentration-time curve from zero to infinity.

SECONDARY OUTCOMES:
Tmax | 0-72 hours post dose
  time to reach maximum plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Raeefuddin Ahmed, MD, Study Director — Abbott
Locations (1):
- Center for Bioequivalence Studies and Clinical Research (CBSCR) ICCBS, University of Karachi, Karachi, Sindh, Pakistan